CLINICAL TRIAL: NCT03662802
Title: Development of a Novel Convolution Neural Network for Arrhythmia Classification for Shockable Cardiac Rhythms
Brief Title: Development of a Novel Convolution Neural Network for Arrhythmia Classification
Acronym: AI-ECG
Status: Completed | Type: Observational
Sponsor: Scripps Clinic (Other)
Responsible Party: Principal Investigator, Sanjeev Bhavnani MD, Principal Investigator - Healthcare Innovation, Scripps Clinic
Organization: Scripps Health (Other)
Other Study IDs: 027527
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Arrhythmias, Cardiac; Cardiac Arrest; Cardiac Arrythmias
Keywords: artificial intelligence; machine learning; neural network; cardiac arrhythmia; ECG; EKG
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECG Data: Coded data including; wavelengths, amplitude, intervals, timing, frequence
  Interventions: Other: Neural Network Classifier

INTERVENTIONS:
Other: Neural Network Classifier — The convolutional neural network is configured to receive an electrocardiogram segment as an input and to generate an output indicative of whether the received electrocardiogram segment represents a cardiac arrhythmia. No specific features of the electrocardiogram are identified to the convolutional neural network, and the received electrocardiogram segment is not filtered, transformed, or processed prior to reception by the algorithm. The algorithm is trained in a similar manner - the electrocardiogram segments are the sole input to the convolutional neural network.

SUMMARY:
Identifying the correct arrhythmia at the time of a clinic event including cardiac arrest is of high priority to patients, healthcare organizations, and to public health. Recent developments in artificial intelligence and machine learning are providing new opportunities to rapidly and accurately diagnose cardiac arrhythmias and for how new mobile health and cardiac telemetry devices are used in patient care. The current investigation aims to validate a new artificial intelligence statistical approach called 'convolution neural network classifier' and its performance to different arrhythmias diagnosed on 12-lead ECGs and single-lead Holter/event monitoring. These arrhythmias include; atrial fibrillation, supraventricular tachycardia, AV-block, asystole, ventricular tachycardia and ventricular fibrillation, and will be benchmarked to the American Heart Association performance criteria (95% one-sided confidence interval of 67-92% based on arrhythmia type). In order to do so, the study approach is to create a large ECG database of de-identified raw ECG data, and to train the neural network on the ECG data in order to improve the diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* All ECG data compiled from 12-lead ECG, single, and multiple lead databases

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals undergoing a 12-lead ECG or Holter/Event monitoring
Sampling Method: Non-Probability Sample
Enrollment: 25458 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy | 1 YEAR
  American Heart Association ECG Performance Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Bhavnani, MD, Principal Investigator — Scripps Clinic Medical Group
Locations (1):
- Scripps Clinic, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson KW, Torres Soto J, Glicksberg BS, Shameer K, Miotto R, Ali M, Ashley E, Dudley JT. Artificial Intelligence in Cardiology. J Am Coll Cardiol. 2018 Jun 12;71(23):2668-2679. doi: 10.1016/j.jacc.2018.03.521. PMID 29880128
- [Background] Kiranyaz S, Ince T, Gabbouj M. Real-Time Patient-Specific ECG Classification by 1-D Convolutional Neural Networks. IEEE Trans Biomed Eng. 2016 Mar;63(3):664-75. doi: 10.1109/TBME.2015.2468589. Epub 2015 Aug 14. PMID 26285054
- [Result] Bhavnani SP, Parakh K, Atreja A, Druz R, Graham GN, Hayek SS, Krumholz HM, Maddox TM, Majmudar MD, Rumsfeld JS, Shah BR. 2017 Roadmap for Innovation-ACC Health Policy Statement on Healthcare Transformation in the Era of Digital Health, Big Data, and Precision Health: A Report of the American College of Cardiology Task Force on Health Policy Statements and Systems of Care. J Am Coll Cardiol. 2017 Nov 28;70(21):2696-2718. doi: 10.1016/j.jacc.2017.10.018. No abstract available. PMID 29169478
- [Result] Bhavnani SP, Narula J, Sengupta PP. Mobile technology and the digitization of healthcare. Eur Heart J. 2016 May 7;37(18):1428-38. doi: 10.1093/eurheartj/ehv770. Epub 2016 Feb 11. PMID 26873093
- [Result] Vandendriessche B, Abas M, Dick TE, Loparo KA, Jacono FJ. A Framework for Patient State Tracking by Classifying Multiscalar Physiologic Waveform Features. IEEE Trans Biomed Eng. 2017 Dec;64(12):2890-2900. doi: 10.1109/TBME.2017.2684244. Epub 2017 Mar 17. PMID 28328498
- [Result] Arvanaghi R, Daneshvar S, Seyedarabi H, Goshvarpour A. Fusion of ECG and ABP signals based on wavelet transform for cardiac arrhythmias classification. Comput Methods Programs Biomed. 2017 Nov;151:71-78. doi: 10.1016/j.cmpb.2017.08.013. Epub 2017 Aug 24. PMID 28947007
- [Result] Figuera C, Irusta U, Morgado E, Aramendi E, Ayala U, Wik L, Kramer-Johansen J, Eftestol T, Alonso-Atienza F. Machine Learning Techniques for the Detection of Shockable Rhythms in Automated External Defibrillators. PLoS One. 2016 Jul 21;11(7):e0159654. doi: 10.1371/journal.pone.0159654. eCollection 2016. PMID 27441719
- [Result] Li Q, Rajagopalan C, Clifford GD. Ventricular fibrillation and tachycardia classification using a machine learning approach. IEEE Trans Biomed Eng. 2014 Jun;61(6):1607-13. doi: 10.1109/TBME.2013.2275000. Epub 2013 Jul 26. PMID 23899591
- [Result] Lyon A, Minchole A, Martinez JP, Laguna P, Rodriguez B. Computational techniques for ECG analysis and interpretation in light of their contribution to medical advances. J R Soc Interface. 2018 Jan;15(138):20170821. doi: 10.1098/rsif.2017.0821. PMID 29321268
- [Result] Mjahad A, Rosado-Munoz A, Bataller-Mompean M, Frances-Villora JV, Guerrero-Martinez JF. Ventricular Fibrillation and Tachycardia detection from surface ECG using time-frequency representation images as input dataset for machine learning. Comput Methods Programs Biomed. 2017 Apr;141:119-127. doi: 10.1016/j.cmpb.2017.02.010. Epub 2017 Feb 10. PMID 28241963
- [Result] Xiong Z, Nash MP, Cheng E, Fedorov VV, Stiles MK, Zhao J. ECG signal classification for the detection of cardiac arrhythmias using a convolutional recurrent neural network. Physiol Meas. 2018 Sep 24;39(9):094006. doi: 10.1088/1361-6579/aad9ed. PMID 30102248
- [Result] Fan X, Yao Q, Cai Y, Miao F, Sun F, Li Y. Multiscaled Fusion of Deep Convolutional Neural Networks for Screening Atrial Fibrillation From Single Lead Short ECG Recordings. IEEE J Biomed Health Inform. 2018 Nov;22(6):1744-1753. doi: 10.1109/JBHI.2018.2858789. Epub 2018 Aug 7. PMID 30106699
- [Result] Warrick PA, Nabhan Homsi M. Ensembling convolutional and long short-term memory networks for electrocardiogram arrhythmia detection. Physiol Meas. 2018 Oct 30;39(11):114002. doi: 10.1088/1361-6579/aad386. PMID 30010088
- [Derived] Shen CP, Freed BC, Walter DP, Perry JC, Barakat AF, Elashery ARA, Shah KS, Kutty S, McGillion M, Ng FS, Khedraki R, Nayak KR, Rogers JD, Bhavnani SP. Convolution Neural Network Algorithm for Shockable Arrhythmia Classification Within a Digitally Connected Automated External Defibrillator. J Am Heart Assoc. 2023 Apr 18;12(8):e026974. doi: 10.1161/JAHA.122.026974. Epub 2023 Mar 21. PMID 36942628